CLINICAL TRIAL: NCT06211270
Title: Food and Resources Expanded to Support Health and Type 2 Diabetes (FRESH-T2D)
Brief Title: Food and Resources Expanded to Support Health and Type 2 Diabetes
Acronym: FRESH
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: El Rio Community Health Center (Other); Arizona State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01DK132300-01A1 (NIH)
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Randomized wait-list controlled pilot study using a convergent mixed methods approach
Who Masked: Outcomes Assessor
Masking Description: Data collectors are blinded to participant's study arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): FRESH-T2D Intervention consisting of bimonthly food, recipes, and diabetes self-management resources + 4 meetings with Registered Dietitian Nutritionists x 6 months duration
  Interventions: Behavioral: FRESH
- Wait-Listed Control (Other): Standard of Care for El Rio Community Health Center persons with type 2 diabetes.
  Interventions: Behavioral: FRESH

INTERVENTIONS:
Behavioral: FRESH — FRESH-T2D Intervention consisting of bimonthly food, recipes, and diabetes self-management resources + 4 meetings with Registered Dietitian Nutritionists x 6 months duration

SUMMARY:
Food insecurity, poor nutrition, and economic disadvantage are critical social determinants of health that contribute to disparities in type 2 diabetes mellitus (T2DM), a serious diet-sensitive chronic disease affecting more than 20% of food insecure adults. There is a demonstrable need for food-focused interventions to address the diet quality of persons with, or at risk of, T2DM. Completion of the pilot study will produce recruitment, retention, adherence, and cost data for a future definitive randomized controlled clinical trial, bringing us closer to the long-term goal of a tested, efficacious model of diabetes care coordinated across Federally Qualified Health Centers and food bank networks.

DETAILED DESCRIPTION:
In 2020, more than 38.5 million (10.5%) U.S. households were without reliable access to sufficient quantities of affordable, nutritious food due to limited money or other resources. Food insecurity, poor nutrition, and economic disadvantage are critical social determinants of health that contribute to disparities in type 2 diabetes mellitus (T2DM), a serious diet-sensitive chronic disease affecting more than 20% of food insecure adults. Coping strategies favor inexpensive, ultra-processed foods that substantially diminish diet quality and are associated with increased incidence and severity of T2DM, including poorer glycemic control and excess body weight. Given that numerous social factors and systems contribute to and perpetuate food insecurity and poor diabetes outcomes, there is a demonstrable need for multilevel (individual, household, community) food-focused interventions to effectively and sustainably address the diet quality of persons with, or at risk of, T2DM. To date, no studies have rigorously tested whether intervention programs explicitly designed to improve both food and nutrition security of low-income persons with T2DM are feasibly delivered by personnel at a Federally Qualified Health Center (FQHC), acceptable to patients seeking care in their medical home, or are capable of producing clinically relevant changes in T2DM endpoints. These are questions will be explored in the proposed randomized wait-list controlled pilot study- Food and Resources Expanded to Support Health and Type 2 Diabetes (FRESH-T2DM)- in which a previously developed food and diabetes self-management education (DSME) intervention (FRESH) will be delivered to 50 adult FQHC patients with T2DM and food insecurity twice monthly, for 6 months. The FRESH intervention consists of bimonthly food provision; a series of recipes that feature FRESH foods; diabetes self-management education (DSME) resources; and four, 30-minute visits with an FQHC Registered Dietitian Nutritionist and Certified Diabetes Educator who will help participants utilize FRESH resources to meet personalized treatment goals. Building upon prior work and existing collaborations with colleagues at El Rio Community Health Center, a Federally Qualified Health Center serving >110,000 underinsured, uninsured patients and the Community Food Bank of Southern Arizona, a regional food bank serving 180,000 Arizonans across 5 counties, the Specific Aims are to: (Specific Aim 1) Assess the feasibility, acceptability, and participant uptake of the FRESH intervention, delivered to 50 food insecure adults with T2DM at their medical home, El Rio Community Health Center, and (Specific Aim 2) Explore changes in blood glucose control, diet quality, food security, diabetes self-care behaviors, and health-related quality of life among participants at 3 and 6 months. Completion of this pilot study -submitted in response to NIDDK PAS-20-160 -will produce data to inform the rationale and design of a future definitive randomized controlled clinical trial, including recruitment, retention, adherence, and cost data. The long-term goal is to produce a tested, efficacious model of coordinated care capable of replication and scaling across other FQHCs and food bank networks.

ELIGIBILITY:
Inclusion Criteria:

* adult (ages 18+); patient at El Rio Community Health Center; fluent in English or Spanish; physician diagnosis of T2DM; food insecure (based on a "yes" answer to the 2-item Hunger Vital Sign food security screening tool used by El Rio to screen patients); stable housing with access to a kitchen; U.S.-based address and telephone number; willingness to participate in all study activities (Section C.6) for the duration of the study (12 months on study, including 6 months of intervention).

Exclusion Criteria:

* diagnosed psychiatric disturbances or mental illness; physical limitations or medical conditions restricting ad libitum food intake (e.g., dysphagia); inability to read and write; no home phone or home address; not able to speak and read English or Spanish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-09-13 (Actual); Primary Completion 2025-10-24 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Acceptability Aim 1 | 6 months (post-intervention)
  How participants and those involved in implementing the program react to the intervention, assessed via qualitative in-depth interviews. Satisfaction with foods and resources, suggestions for improvement, perceived usefulness will be explored.
Demand | 6 months (post-intervention)
  Intervention uptake (relevance of foods/resources/services provided, promoters and barriers to participation in the intervention, degree to which participants report using the intervention resources to influence T2DM, "fit" with daily life, cultural congruence) will be explored in brief surveys and qualitative in-depth interviews.
Implementation | 3- and 6 months (post-intervention), and 12 months (follow-up)
  The extent, likelihood, and manner in which the intervention is implemented as planned, including participant recruitment and retention rates and ease/burden associated with data collection methods will be estimated from research team logs, and qualitative in-depth interviews. Retention rate will be calculated at study end (12 months).
Practicality | Throughout the intervention, and at 6 months (post-intervention)
  Adherence(# of boxes received, resources utilized, and RDN/CDE visits completed), will be calculated from research team logs. Costs, burden and benefit the participants and the FQHC will be evaluated using a bottom-up micro-costing approach - for participants, this will include time and resources spent in travel, and services, equipment, and food needed to meet program recommendations; for the FQHC, this includes direct medical and non-medical costs including personnel gross hourly salaries, intervention material costs (in partnership with the Food Bank), and overhead costs related to use of facilities for prevention services will be tracked and analyzed in partnership with FQHC data team members; 5) any adaptation or modifications of the intervention by the FQHC to accommodate patients and organization.
Adaptation | 6 months (post-intervention)
  Any modifications of the intervention by the FQHC to accommodate patients and organizational requirements and context will be explored through qualitative in-depth interviews with FQHC and Food Bank personnel.
Expansion | 6 months (post-intervention)
  Potential for sustainability of the program at the FQHC, and expansion of the intervention across other FQHCs, and any positive or negative effects on the organization will be explored through qualitative in-depth interviews with FQHC personnel.
Integration | 6 months (post-intervention)
  Integration of the FRESH intervention with provider care plans for patients, a systems-level change that would allow the program to be a reimbursable treatment, will be explored through qualitative in-depth interviews with FQHC personnel.

SECONDARY OUTCOMES:
Demographics and Social Determinants of Health | Baseline, 3- and 6 months (post-intervention)
  Self-reported using the Protocol for Responding to and Assessing Patients' Assets, Risks, and Experiences (PRAPARE) Questionnaire, a screening tool used by Federally Qualified Health Centers to better understand social determinants of health.
Glycated hemoglobin (HbA1c) | Baseline, 3- and 6 months (post-intervention)
  HbA1c is an established metric for long-term monitoring of blood glucose control in persons with T2DM. HbA1c will be collected by the research team using portable (point-of-care) capillary-based technology (Siemens Diagnostics DCA HbA1C analyzer).
Dietary intake and diet quality | Baseline, 3- and 6 months (post-intervention)
  Typical intake will be assessed using three, non-consecutive (2 weekdays, 1 weekend day), interviewer-administered 24-hour dietary recalls at each measurement time point, conducted telephonically by trained nutritionists and entered into the Nutrient Data System for Research (Minneapolis, MN, v. 2012) From these data, diet quality and its components (total vegetables, whole fruit, whole grains, plant, animal, and seafood proteins, fatty acids, sodium, sugar, and refined grains) will be calculated using the Healthy Eating Index (HEI-2015), a valid and reliable measure of diet quality designed to assess the degree to which an individual's intake conforms to dietary recommendations.
Food security | Baseline, 3- and 6 months (post-intervention)
  USDA 6-item Food Security Questionnaire. Eight additional items from the Current Population Survey Food Security Supplement will allow us to assess food access, expenditures, use of food assistance programs, and other ways of coping with food insecurity.
Perceived adherence to diabetes self-care behaviors | Baseline, 3- and 6 months (post-intervention)
  The Self Care Inventory-Revised (SCI-R) a brief, psychometrically sound measure of patient perceptions of adherence to recommended diabetes self-care behaviors. The SCI-R accommodates various treatment regimens across individuals, while evaluating individuals' perceptions of how well they adhere to their treatment plans.
Health-related quality of life | Baseline, 3- and 6 months (post-intervention)
  The CDC's 4-item Healthy Days Measure asks participants about recent pain, depression, anxiety, sleeplessness, vitality, and the cause, duration, and severity of a current activity limitation an individual may have in their life.
Height | Baseline, 3- and 6 months (post-intervention)
  Height will be measured using a calibrated Seca 213 Portable Stadiometer. All measures will be completed in duplicate, and the average of the two measures will be used.
Body weight | Body weight will be measured using a calibrated Cardinal Detecto 758C Weight Indicator scale. All measures will be completed in duplicate, and the average of the two measures will be used.
  Baseline, 3- and 6 months (post-intervention)
Body Mass Index | Baseline, 3- and 6 months (post-intervention)
  Adult BMI will be categorized using international classifications of BMI (normal weight, 18-24.9 kg/m2; overweight, 25-29.9 kg/m2; obesity, >30 kg/m2).

CONTACTS AND LOCATIONS:
Locations (1):
- El Rio Community Health Center, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
Any publications and presentations that authored by the study team will identify where the data will be available and how to access the data, as well as acknowledge the repository and funding source in any publications and presentations. The study team will explore the use of an NIH-funded repository, which will have policies and procedures in place to provide data access to qualified researchers, fully consistent with NIH data sharing policies and applicable laws and regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After the study has concluded in January 2026.
Access Criteria: A resource sharing plan is not required by the NIH for applications requesting <$500,000 in direct costs for any budget period, nor does the NIDDK require a resource sharing plan under the PAS-20-160 funding mechanism. However, in support of research transparency, rigor, and reproducibility, the study investigators will support requests for access to pilot and feasibility data from qualified scientists for specific analyses.